CLINICAL TRIAL: NCT05170074
Title: National, Multicentre Observational Study on Surgical Reconstruction of the Anterior and Apical Compartment of the Pelvic Floor With a Single-incision, Fixation-free Self-Retaining Support Implant (SRS Implant)
Brief Title: Post-market Clinical Follow-up of the SRS Implant
Status: Active, not recruiting | Type: Observational
Sponsor: pfm medical gmbh (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF study SRS implant
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: SRS Implant; Quality of Life; Pelvic Organ Prolapse; Surgical Reconstruction
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SRS implant: Surgical reconstruction of the anterior and apical compartment of the pelvic floor with an SRS implant

SUMMARY:
National, multicentre observational study on surgical reconstruction of the anterior and apical compartment of the pelvic floor with an SRS implant

DETAILED DESCRIPTION:
National, multicentre, prospective observational study on surgical reconstruction of the anterior and apical compartment in seven clinical centres in Germany to obtain post-market information on the SRS implant with a follow-up of 24 months. Patient reported satisfaction (measured by P QoL, Prolapse Quality of Life Questionnaire), anatomic outcome (measured by the POP-Q, Pelvic Organ Prolapse Quantification system) and the rate of complications (measured by adverse events during the study period) are focused.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a symptomatic anterior vaginal wall prolapse with/without apex/uterine prolapse ≥ stage II (according to POP-Q system). This applies to primary as well as recurrent intervention.
2. Age ≥ 21 years.
3. Patient is mentally able to understand the nature, aims, or possible consequences of the PMCF study.
4. Patient information has been provided and written consent exists.

Exclusion Criteria:

1. Contraindications according to the manufacturer's instructions for use.
2. Patient with previous urogynaecological surgeries with alloplastic material.
3. Patient with radiological treatment in the pelvic floor.
4. Patient is institutionalised by court or official order (MPDG §27).
5. Participation in another interventional study concerning pelvic floor reconstruction.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a symptomatic anterior vaginal wall prolapse with/without apex/uterine prolapse ≥ stage II (according to POP-Q system), transvaginal SRS implantation for pelvic organ prolapse surgery
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient´s Quality of Life | 12 months
  Evaluation of changes in quality of life twelve months after implantation of the SRS implant compared to baseline. Quality of Life was assessed by the P-QOL (Prolapse Quality of Life Questionnaire). The P-QOL yields a domain score in the range from zero to 100, wheras a score of zero is the best.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cadenbach-Blome, Dr. med., Principal Investigator — Asklepios Klinik Altona
Locations (7):
- Germany (7):
  - Heilig Geist-Hospital, Bensheim, Hesse
  - Universitätsklinikum Augsburg, Augsburg
  - Evangelisches Krankenhaus Hagen-Haspe, Hagen
  - Asklepios Klinik Altona, Hamburg
  - Städtisches Krankenhaus Kiel, Kiel
  - Marienhaus Klinikum Hetzelstift Neustadt/Weinstraße, Neustadt
  - Klinikum Oberlausitzer Bergland gGmbH, Zittau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy G, Padoa A, Marcus N, Beck A, Fekete Z, Cervigni M. Anchorless implant for the treatment of advanced anterior and apical vaginal prolapse - Medium term follow up. Eur J Obstet Gynecol Reprod Biol. 2020 Mar;246:55-59. doi: 10.1016/j.ejogrb.2020.01.005. Epub 2020 Jan 9. PMID 31954369
- [Background] Levy G, Padoa A, Fekete Z, Bartfai G, Pajor L, Cervigni M. Self-retaining support implant: an anchorless system for the treatment of pelvic organ prolapse-2-year follow-up. Int Urogynecol J. 2018 May;29(5):709-714. doi: 10.1007/s00192-017-3415-3. Epub 2017 Jul 14. PMID 28710613
- See also: Homepage Manufacturer with information on the investigational product — https://lyramedical.com/product/
- See also: Homepage Sponsor with information on the investigational product — https://www.pfmmedical.de/produkte/gynaekologie-senologie/netzimplantate-beckenbodenchirurgie/srs-implantat-ankerloses-single-incision-system,26056/